CLINICAL TRIAL: NCT00020371
Title: Phase I Study of BMS-247550 in Patients With Refractory Neoplasms
Brief Title: BMS-247550 in Treating Patients With Cancers That Have Not Responded to Previous Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068319; NCI-00-C-0224; NCI-550; NCT00006317 (obsolete NCT alias)
Record Dates: First submitted 2007-03-02; First posted 2007-03-06 (Estimated); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific; Neutropenia
Keywords: adult solid tumor; bone marrow suppression; cancer; cancer-related problem/condition; neutropenia; solid tumor; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Neutropenia; Neoplasms | interventions — ixabepilone; Filgrastim

INTERVENTIONS:
Drug: BMS-247550
Drug: filgrastim

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of BMS-247550 in treating patients who have cancers that have not responded to previous therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose, dose-limiting toxic effects, and recommended phase II dose of BMS-247550 in patients with refractory neoplasms.

II. Evaluate the pharmacokinetics and pharmacodynamics of this drug in these patients.

III. Determine the occurrence of response in patients treated with this drug.

PROTOCOL OUTLINE: This is a dose-escalation study. Patients receive BMS-247550 IV over 1 hour on days 1-5. Treatment continues every 3 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 1-6 patients receive escalating doses of BMS-247550 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 6 patients experience dose-limiting toxicity (DLT). Once the MTD is determined, additional patients are accrued to receive BMS-247550 at the recommended phase II dose.

If neutropenia is identified as the DLT, a second dose escalation is performed to identify the MTD of BMS-247550 with the addition of filgrastim (G-CSF) in cohorts as above. Patients receive fixed-dose G-CSF 72 hours after final BMS-247550 dose, and continuing until blood levels return to normal.

PROJECTED ACCRUAL:

A total of 45 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Histologically or cytologically confirmed neoplasm refractory to standard therapy or for which no standard therapy exists No CNS malignancy --Prior/Concurrent Therapy-- Biologic therapy: At least 4 months since prior myeloablative chemotherapy followed by bone marrow or stem cell rescue Chemotherapy: See Biologic therapy At least 4 weeks since prior chemotherapy (6 weeks for prior nitrosoureas or mitomycin) Endocrine therapy: At least 2 weeks since prior hormonal therapy for breast cancer At least 4 weeks since prior hormonal therapy for prostate cancer Radiotherapy: At least 4 weeks since prior radiotherapy No prior craniospinal irradiation, total body irradiation, or radiation to more than half of pelvis Surgery: Not specified Other: No other concurrent investigational drugs --Patient Characteristics-- Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 3 months Hematopoietic: Platelet count at least 100,000/mm3 Absolute granulocyte count at least 1,500/mm3 Hepatic: SGOT/SGPT no greater than 2.5 times normal Bilirubin no greater than 1.5 times normal (no greater than 3 times normal if evidence of Gilbert's disease) Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 50 mL/min Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 2 months after study No other nonmalignant systemic disease or serious medical illness No active uncontrolled infection HIV negative

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2000-09

CONTACTS AND LOCATIONS:
Overall Officials: Jame Abraham, Study Chair — National Cancer Institute (NCI)
Locations (1):
- Medicine Branch, Bethesda, Maryland, United States